CLINICAL TRIAL: NCT00601237
Title: Text Messaging for Abstinence and HIV Risk Prevention: The 411 on Safe Text
Brief Title: Effectiveness of a Cell Phone-Based Program for Abstinence and HIV Risk Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-0463; R21MH083318 (NIH); COMIRB 07-0463; DAHBR 9A-ASPA
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: HIV Infections
Keywords: HIV Prevention; Mobile Phone; Technology-Based Intervention; HIV; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Participants will receive HIV-related text messages
  Interventions: Behavioral: HIV-related text messaging
- B (Active Comparator): Participants will receive nutrition-related text messages
  Interventions: Behavioral: Nutrition-related text messaging
- C (No Intervention): Participants will attend a 90-minute focus group to develop messages for the cell-phone program

INTERVENTIONS:
Behavioral: HIV-related text messaging — Participants will receive up to 90 text messages related to abstinence, monogamy, and condom use over 3 months.
  Arms: A
Behavioral: Nutrition-related text messaging — Participants will receive up to 30 text messages about nutrition and healthy eating over 3 months.
  Arms: B

SUMMARY:
This study will develop and test the effectiveness of a cell phone-based text messaging program to encourage abstinence, monogamy, or condom use among black urban males in Philadelphia, Pennsylvania.

DETAILED DESCRIPTION:
Sexually transmitted diseases (STDs), including HIV infections, are most commonly spread through unprotected sexual intercourse. STDs are a primary health issue, especially among young ethnic minorities in the United States. The rate of STDs is significantly greater in urban areas where ethnic minorities, particularly African-American males, are commonly represented. Despite this information, safe sexual practices, including correct condom use, are not commonly followed among minority males. It is believed that educational outreach designed to motivate and inform on the correct use of condoms will be effective in encouraging safer sex practices. A cell phone-based text messaging program designed to promote safer sex practices may provide an effective and easy means of delivery of treatment. This study will develop and test the effectiveness of a cell phone-based text messaging program to sustain abstinence, monogamy, or condom use among black urban males in Philadelphia, Pennsylvania.

Participation in this study will be divided into two phases. In the first study phase, participants will partake in a 90-minute focus group to help develop text message content and plans for treatment delivery. The next study phase will be a pilot test of the program developed in the first phase. Participants will be assigned to receive text messages concerning either HIV prevention or general nutrition. Participants receiving the HIV prevention text messages will be sent up to 90 text messages related to abstinence, monogamy, and condom use over a 3-month period. Participants will also be able to join interactive phone activities related to HIV. Participants receiving the nutritional text messages will be sent up to 30 messages about nutrition and healthy eating over the same period of time. Participants will complete telephone surveys at baseline and Months 3 and 6. The surveys will assess measures of abstinence, monogamy and condom use attitudes, norms, self-efficacy, and risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Philadelphia
* Self-identified black or African American
* English-speaking
* Cell phone user

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2008-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Condom use | Measured at baseline and Months 3 and 6
Abstinence | Measured at baseline and Months 3 and 6
Monogamy | Measured at baseline and Months 3 and 6

SECONDARY OUTCOMES:
Attitudes, norms, self-efficacy, and intentions to remain abstinent, remain monogamous, or use condoms | Measured at baseline and Months 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Sheana Bull, PhD, Principal Investigator — University of Colorado at Denver and Health Sciences
Locations (1):
- Motivational Educational Entertainment (MEE) Productions, Philadelphia, Pennsylvania, United States